CLINICAL TRIAL: NCT01343940
Title: Project Dulce: Developmental Understanding and Legal Collaboration for Everyone
Brief Title: Strengthening Families and Reducing Risk Thru Developmental and Legal Collaboration
Acronym: dulce
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Center for the Study of Social Policy (Unknown)
Responsible Party: Principal Investigator, Robert Sege, HRIA Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-29958
Record Dates: First submitted 2011-03-16; First posted 2011-04-28 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Parenting; Child Rearing; Child Abuse; Child Neglect; Child Development
Keywords: RCT; randomized block repeated measures design; efficacy trial; high risk population

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dulce family partner intervention (Experimental): Participating families are assigned to a legal/developmental specialist who joins health care team during well-child visits and home visits. The specialist (a "Dulce family partner") supports parent around child development issues, addresses unmet basic needs (e.g., housing, utilities, food, etc.), and makes referral to existing agencies and services.
  Interventions: Behavioral: Project dulce
- Safety intervention (Active Comparator): Participating family is assigned a safety specialist who will provide the parent with guidance, equipment and instruction to reduce risk of newborn injury during transport (car seat) and while sleeping (Pack-and-Play).
  Interventions: Behavioral: Safety intervention

INTERVENTIONS:
Behavioral: Project dulce — Participating families are assigned to a legal/developmental specialist who joins health care team during well-child visits and home visits. The specialist (a "Dulce family partner") supports parent around child development issues, addresses unmet basic needs (e.g., housing, utilities, food, etc.), and makes referral to existing agencies and services. Specialist meets with family during all routine well-child visits scheduled in primary care between birth and 6 months (1-mo, 2-mo, 4-mo, 6-mo). Parent may meet with specialist before or after scheduled appointment, and may request a home visit. Specialist will be available by phone for consultation.
  Other Names: dulce; dulce family partner
  Arms: Dulce family partner intervention
Behavioral: Safety intervention — Participating family is assigned a safety specialist. Meeting with the safety specialist will occur before or after a routine well-child visit or at a separately agreed upon time. The specialist will discuss infant injury risks associated with transportation and sleep. The specialist will provide safety equipment (car seat and pack-and-play) and instruct the parent in their proper use.
  Arms: Safety intervention

SUMMARY:
Project Dulce is designed to test a new approach to delivering family support, in the context of the primary care medical home. The target population to be served is infants between birth and 6 months old and their families who receive primary care at Boston Medical Center. A dulce family partner will reach infants and families through their routine health care visits during their first six months of life and provide them with support for unmet legal needs, screen infants for developmental problems, screen families for mental health problems, and improve families' knowledge of child development. The control group will receive training on safe sleep and safe transportation for their newborn.

DETAILED DESCRIPTION:
Subjects for project dulce will be recruited from parents who receive their newborn child's primary pediatric care from Boston Medical Center's Pediatric Primary Care Clinic. Subjects will be randomized to receive the study intervention or the control.

Project dulce will provide a family partner to parents of infants up to six months of age. The dulce family partner (DFP) will be trained using the Healthy Steps model, an evidence-based approach to support parent understanding of child development, and by Medical Legal Partnership|Boston to identify legal and social needs that may affect a child's health and development. The dulce family partner will reach infants and families through their routine health care visits during their first six months of life and provide them with support for unmet legal needs, screen infants for developmental problems, screen families for mental health problems, and improve families' knowledge of child development. Families will meet with the DFP at the initial visit, at their subsequent routine healthcare maintenance visits, and during home visits if they wish.

Families in the control group will receive safety education from a trained staff member on safe sleep and safe transportation, at two of their baby's routine well-child visits between 1 and 6 months of age.

Subjects will answer two sets of standard survey questions before and after intervention / control. The infant's electronic medical record will be reviewed up to the first year. This study will test whether the project dulce intervention promotes positive outcomes for children and families, and reduces risks and adverse outcomes. The results of this rigorous program evaluation may be used to support dissemination of project dulce to other primary care sites throughout the country.

PROJECT GOALS 1. Assess whether the highly-structured dulce intervention results in: improved individual and family strengths, reduced risks, and decreased likelihood of child maltreatment. 2. Provide system-level information to assess the costs, resource needs, barriers, and benefits that come from implementing the dulce model within a patient-centered medical home. 3. In addition to the project's research goals, we will collect aggregated Child Protective Service (CPS) community-wide data regarding childhood injury and maltreatment, as is requested by funder.

ELIGIBILITY:
Inclusion Criteria:

* The patient family must include an infant, or infants for families with multiples, born 10 weeks or less prior to recruitment.
* The newborn(s) must be healthy, having been born without known defects or complications that would require early hospitalization.
* The infant must have been discharged from hospital within one week.
* At the time of recruitment, the parent/guardian will have communicated their intent to obtain their newborn infant's primary pediatric care through Boston Medical Center's (BMC's) Primary Pediatric Care Clinic (PPCC).
* The child's parent/guardian must be able to engage in an informed consent process conducted in English or Spanish.
* The child's parent/guardian must be able to complete a questionnaire and/or interview (with or without assistance) in English or Spanish.

Exclusion Criteria:

* The participating parent/guardian is under 18 years of age. As SOC at BMC, mothers under the age of 18 are seen in the The Teen and Tot Program (TTP), a specialized program located within BMC's Adolescent Center.
* The parent/guardian is unable to participate in required data collection activities in the study languages, even with assistance.
* The child/family's physician believes that participation in the evaluation would adversely affect the child/family's health or well being or the ongoing delivery of health care services. Decision will be made based on the physician's clinical judgment. All physicians have the opportunity to opt their patients out.
* The family is already receiving services from another family partner program such as Project RISE, Healthy Steps, etc. through the BMC primary care center.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of child maltreatment protective factors available to caregiver at 6 months, as measured on the Quality Improvement Center on Early Childhood (QIC) "Caregivers Assessment of Protective Factors" | t1 (Baseline): at recruitment, prior to intervention; and t2: 6 months later
  Paper-and-pencil questionnaire completed by child's caregiver
Change from baseline in number and amount of income supports available to and accessed by caregiver at 6 months, as measured on the Quality Improvement Center on Early Childhood (QIC) "Self-Report Family Inventory" + supplementary questions on $ value | t1 (Baseline): at recruitment, prior to intervention; and t2: 6 months later
  Paper-and-pencil questionnaire completed by child's caregiver
Change from baseline in social capital available to caregiver at 6 months, as measured on the Quality Improvement Center on Early Childhood (QIC) "Social Network Grid" | t1 (Baseline): at recruitment, prior to intervention; and t2: 6 months later
  Paper-and-pencil questionnaire completed by child's caregiver working with reasearch interviewer. Adapted from: Tracy, EM & Whittaker, JK (1990). The Social Network Map: Assessing social support in clinical social work practice. Families in Society, 71(8), 461-470.
Change from baseline in parental stress at 6 months, as measured by the "Parenting Stress Index (PSI) - long form" | t1 (Baseline): at recruitment, prior to intervention; and t2: 6 months later
  Paper-and-pencil instrument completed by child's caregiver
Change from baseline in parenting and child-rearing attitudes of child's caregiver at 6 months, as measured on the "Adult-Adolescent Parenting Inventory(AAPI-2)" | t1 (Baseline): at recruitment, prior to intervention; and t2: 6 months later
  Paper-and-pencil instrument completed by child's caregiver; 40 Likert-type items.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Sege, MD, PhD, Principal Investigator — Boston University; Edward De Vos, EdD, Study Director — William James College
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sege R, Preer G, Morton SJ, Cabral H, Morakinyo O, Lee V, Abreu C, De Vos E, Kaplan-Sanoff M. Medical-Legal Strategies to Improve Infant Health Care: A Randomized Trial. Pediatrics. 2015 Jul;136(1):97-106. doi: 10.1542/peds.2014-2955. Epub 2015 Jun 1. PMID 26034248
- [Result] Sege R., Kaplan-Sanoff M., Morton S., Velasco-Hodgson M.C., Preer G., Morakinyo G., De Vos E., Krathen J. Project DULCE: Strengthening families through enhanced primary care. The Journal of Zero to Three. Vol 35(1):10-18, September 2014.